CLINICAL TRIAL: NCT03914716
Title: Radiogenomics: Personalized Imaging of Arthropathy in Boys With Hemophilia in China
Brief Title: Imaging of Arthropathy in Boys With Hemophilia in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andrea Doria (Other)
Collaborators: Beijing Children's Hospital, Baxalta US Inc. (Unknown)
Responsible Party: Sponsor-Investigator, Andrea Doria, Radiologist, Senior Scientist, Research Director, Department of Diagnostic Imaging, The Hospital for Sick Children
Organization: The Hospital for Sick Children (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1000058500
Record Dates: First submitted 2019-02-19; First posted 2019-04-16 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Hemophilia
Keywords: Hemophilia; Radiogenomics; Arthropathy
MeSH Terms: conditions — Hemophilia A; Joint Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Study group — Subjects will have physical, imaging examinations and provide samples for biological markers

SUMMARY:
Hemophilia is a genetic condition characterized by marked phenotypic heterogeneity. Bleeding into a joint is the single most important risk factor for the development of hemophilic arthropathy (HA). It is thought that clinical and imaging manifestations of HA are at least partially attributable to genetic polymorphisms unrelated to the hemophilia genotype. Identifying and characterizing biologic factors that could explain differences in susceptibility to joint degeneration of patients with hemophilia would help stratify patients according to the risk of degeneration of their joints and develop personalized therapeutic and prophylactic strategies. This study is conducted in China.

DETAILED DESCRIPTION:
This will be a 3-year prospective cohort study conducted in a single centre (Beijing Children's Hospital, BCH, China) with a 2-year follow-up of patients Index joints (ankles, elbows and knees) of young Chinese boys with hemophilia A will be evaluated as follows: physical examination every 6 months using the Hemophilia Joint Health Score [HJHS], ultrasound imaging (gray-scale and color Doppler ultrasound [US]), and by laboratory (serum) at baseline, at 6, and 24 months. Magnetic resonance imaging (MRI) scans of index joints will be obtained at baseline, and 24 months. Features that will be captured either quantitatively or semantically in the imaging scans will be aggregated to generate "imaging phenotypes" which will be associated with clusters of co-expressed genes (metagenes) and clinical data.

ELIGIBILITY:
Inclusion Criteria:

* Hemophilia A with baseline FVIII levels of <2%
* Clinical history of ≥ 50 exposure days to FVIII prior to the study start.
* On-demand treatment, prophylaxis FVIII infusions or treatment with plasma-derived products for >3 months prior to enrollment into the study.

Exclusion Criteria:

* History of FVIII inhibitor (titer >0.6 Bethesda Units [BU])
* Chronic renal failure (serum creatinine >2.0 mg /dL).
* Chronic liver disease (alanine aminotransferase [ALT] >200 U/L).
* Clinically documented immunodeficiency.
* Anticipation of need for major surgery during the study period.
* Association of diseases known to mimic or cause joint diseases such as symptomatic human immunodeficiency virus (HIV) infection, juvenile idiopathic arthritis, and metabolic bone diseases.
* Social barriers for participation in the study such as long distance between home and the comprehensive care centre, and documented track record of non-compliance to therapies or participation in clinical studies.
* Neuro-developmental/behavioral problems.
* Contraindications to MR imaging (presence of heart pacemakers, metallic foreign bodies in the eye, aneurysm clips, severe claustrophobia).

Ages: 4 Years to 11 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Annualized total index joint bleeding rates (AJBRs) | Between baseline and 24 months
  AJBRs will be calculated from prospectively collected joint bleeding logs and clinic records.

SECONDARY OUTCOMES:
Number of participants with joint inflammation | At baseline, 6 months and 24 months
  Assessed by ultrasound
Number of participants with joint inflammation | Between baseline and 24 months
  Assessed by MRI of the joints
Number of participants with joint damage | At baseline, 6 months and 24 months
  Assessed by ultrasound
Number of participants with joint damage | Between baseline and 24 months
  Assessed by MRI of the joints
Number of participants with clinical arthropathy | Every 6 months
  Assessed by the Hemophilia Joint Health Score tool (HJHS), version 2.1 - Joint score range: 0 (normal) to 16 (worse outcome).
Presence of inflammatory biomarkers in plasma | At baseline, 6 months and 24 months
  Measured by ELISA (enzyme-linked immunosorbent assay)
Internal MRI-based soft tissue score change | Between baseline and 24 months
  Assessed by the 17-point International Prophylaxis Study Group (IPSG) MRI scale. Score range: 0 to 17 (worse outcome)
Internal MRI-based osteochondral tissue score change | Between baseline and 24 months
  Assessed by the 17-point International Prophylaxis Study Group (IPSG) MRI scale. Score range: 0 to 17 (worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Doria, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Beijing Children's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No